CLINICAL TRIAL: NCT00885872
Title: A 104-week, Open-label, Single-group Study: Rosuvastatin Evaluation of Atherosclerotic Chinese Patients (REACH)
Brief Title: Rosuvastatin Evaluation of Atherosclerotic Chinese Patients (REACH)
Acronym: REACH
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese PLA General Hospital (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Ye Ping/ Director, Chinese PLA General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REACH; D3560L00091 (Other: Astrazeneca)
Record Dates: First submitted 2009-04-21; First posted 2009-04-22 (Estimated); Last update posted 2010-05-27 (Estimated); Status verified 2009-04

CONDITIONS: Hyperlipidemia; Atherosclerosis
MeSH Terms: conditions — Hyperlipidemias; Atherosclerosis | interventions — Rosuvastatin Calcium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treat (Experimental): At visit 2 each eligible subject will be allocated to rosuvastatin. Subjects who reach the criteria at visit 3, dosage of rosuvastatin will be titrated. The subjects will be encouraged to take the study drug at the same time each day for 104 weeks.
  Interventions: Drug: Rosuvastatin (Crestor)

INTERVENTIONS:
Drug: Rosuvastatin (Crestor) — at visit 2 each eligible subject will be allocated to rosuvastatin. study medication wil be taken orally with water once daily, as directed by the study physician. subjects who meet the criteria at visit 3, dosage of rosuvastatin will be titrated.
  Other Names: Crestor

SUMMARY:
This study is to evaluate the effect of rosuvastatin 10-20 mg on carotid atherosclerosis progression in Chinese patients by evaluating the change in the percentage of volume of lipid rich necrotic core (LRNC) using high-resolution magnetic resonance imaging (MRI) after 24-months treatment.

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate the effect of rosuvastatin 10-20 mg on carotid atherosclerosis progression in Chinese patients by evaluating the change in the percentage of volume of lipid rich necrotic core (LRNC) using high-resolution magnetic resonance imaging (MRI) after 24-months treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients between 18 and 75 years of age, inclusive.
2. LDL-C concentration ≥ 100mg/dl (2.6mmol/L), but less than 250mg/dl (6.5mmol/L); and TG ≤ 353mg/dl (4.0mmol/L).
3. New patients in regard to statin therapy.
4. 16%-69% carotid artery stenosis by duplex ultrasound. At least one or more carotid plaques detectable in either the right or left side of the carotid artery 2.4 cm proximal and 2.4 cm distal to the bifurcation. Plaque must be more than 3 mm thick with calcification presenting less than 50% of the plaque area. The plaque must have a LRNC and intact fibrous cap detected by contrast-enhanced MRI (CE MRI).
5. Female patients must agree to use an effective form of birth control throughout the 2-year study treatment period. They must be either documented post-menopausal, physically or surgically incapable of bearing children, or using barrier contraceptive methods. In addition to using contraception, women of childbearing potential must also have a negative serum pregnancy test at Screening.
6. The patients who are willing to be enrolled have to remain on the low cholesterol dietary (refer to Chinese Guideline on Treatment of Dyslipidemia in Adult) for the study duration.
7. The patient must be able to comply with scheduled visits, the treatment plan and all laboratory tests.
8. The patient must provide written voluntary informed consent to participate in the study.

Exclusion Criteria:

1. The patient has liver function tests > 1.5 times the upper limit of normal, serum creatinine > 2.0 mg/dL, GFR < 30 ml/min or has abnormal laboratory values which are deemed clinically significant by the investigator.
2. The patient has severe heart disease, including NYHA III-IV, uncontrolled arrhythmia and acute coronary syndrome. The patient has had a coronary artery bypass graft (CABG), percutaneous coronary intervention (PCI), carotid endarterectomy (CEA), carotid artery stent, or lower extremity revascularization/amputation. The patient had unstable angina or myocardial infarct within 3 months before enrolment.
3. The patient has plans for surgical/endovascular intervention for carotid, coronary and/or peripheral arterial disease during the course of the study.
4. The patient has critical limb ischemia, as evidenced by ischemic rest pain, ulceration, or gangrene.
5. The patient has or is being treated or evaluated for diagnosed tuberculosis. The patient has had a chest x-ray obtained within the last month which shows signs consistent with possible tuberculosis.
6. The patient has a history of malignant neoplasm within the previous 5 years (exception: curable non-melanoma skin malignancies).
7. The patient has a known immunodeficient state (e.g., human immunodeficiency virus) or is being treated with immunosuppressive drugs including cyclosporine.
8. The patient have to take medicines as follow:

   * Hormonal therapy
   * Cyclosporine
   * Other lipid lowering agents: fish oil, garlic essential oil etc.
9. The patient has suffered deep vein thrombosis within the previous 3 months.
10. The patient has suffered brain haemorrhage before the study.
11. The patient has a history of recent alcohol abuse, drug abuse or significant mental illness.
12. The patient has any condition that would prevent the patient from giving voluntary informed consent.
13. The patient has an inability to tolerate oral medication administration.
14. The patient has a known or suspected allergy to the study medication(s) or the class of study medication to be administered.
15. The patient has a known or suspected allergy to MRI contrast agents (e.g., gadolinium).
16. The patient is enrolled or plans to enroll in another clinical drug or device/interventional trial during this study.
17. The patient has any other clinically significant medical condition that, in the opinion of the Investigator, could impact the patient's ability to successfully complete the trial.
18. The patient has the history of myopathy.
19. The patient has the history of epilepsy/seizures.
20. The patient has thyroid stimulating hormone (TSH) > 1.5xULN.
21. The patients has LDL cholesterol > 250mg/dL or total cholesterol > 309 mg/dL or familial hypercholesterolemia.
22. The patient has uncontrolled hypertension, with SBP >160 mmHg and / or DBP >100 mmHg.
23. The patient has uncontrolled hyperglycemia with HbA1c > 9% or diagnosed as DM recently (within 1 month before enrolment)
24. BMI ≥ 30 kg/m2
25. The patient has a pacemaker or other metallic foreign body.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2009-03; Primary Completion 2012-03 (Estimated); Study Completion 2012-03 (Estimated)

PRIMARY OUTCOMES:
Change in the percentage of volume of lipid rich necrotic core (LRNC)using high-resolution MRI | 2 years
  Disease progresson will be determined by the change in the percentage of volume of LRNC measured at 104 weeks (+/-14days) following the initiation of drug treatment in patients with atherosclerotic disease from baseline

SECONDARY OUTCOMES:
change in volume of wall and normalized wall index (NWI) | 2 years
  change in volume of wall and NWI measured at 13 weeks (+/-7days), 52 weeks (+/-7days), and 104 weeks (+/- 7days) following the initiation of drug treatment in patients with atherosclerotic disease from baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Ping Ye, Doctor, Principal Investigator — Chinese PLA General Hospital
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Du R, Cai J, Zhao XQ, Wang QJ, Liu DQ, Leng WX, Gao P, Wu HM, Ma L, Ye P. Early decrease in carotid plaque lipid content as assessed by magnetic resonance imaging during treatment of rosuvastatin. BMC Cardiovasc Disord. 2014 Jul 14;14:83. doi: 10.1186/1471-2261-14-83. PMID 25022285